CLINICAL TRIAL: NCT00171106
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Determine the Effects of Valsartan on Exercise Time in Subjects With Symptomatic Diastolic Heart Failure
Brief Title: Efficacy and Safety of Valsartan Versus Placebo on Exercise Tolerance in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489B2401
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diastolic Dysfunction, Symptomatic Heart Failure
Keywords: diastolic dysfunction; heart failure; exercise tolerance; valsartan
MeSH Terms: conditions — Heart Failure | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
This study will test the effects of valsartan versus placebo on exercise tolerance in patients with symptoms of heart failure

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic diastolic heart failure
* Breathlessness with physical exertion

Exclusion Criteria:

* Uncontrolled hypertension
* Asthma, COPD, or abnormal lung function
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Allergy to valsartan

Other protocol-defined exclusion criteria may apply

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-12; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in baseline exercise test after 15-42 days and 14 weeks

SECONDARY OUTCOMES:
Oxygen consumption during the exercise test
Exercise test blood pressure
Borg score of breathlessness
6-minute walk test at baseline and after 14 weeks
Quality of life assessment at baseline and after 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Parthasarathy HK, Pieske B, Weisskopf M, Andrews CD, Brunel P, Struthers AD, MacDonald TM. A randomized, double-blind, placebo-controlled study to determine the effects of valsartan on exercise time in patients with symptomatic heart failure with preserved ejection fraction. Eur J Heart Fail. 2009 Oct;11(10):980-9. doi: 10.1093/eurjhf/hfp120. PMID 19789402